CLINICAL TRIAL: NCT07165561
Title: Evaluation of an App for Young People With Suicidal Thoughts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2024-0547
Record Dates: First submitted 2025-08-22; First posted 2025-09-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Suicidal Behavior; Suicidal Ideation; Coping Behavior
Keywords: suicidal ideation; adolescents; suicidal behavior; Suicide-Related Coping; e-mental health
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Once the participants and their parents/guardians have given their consent online, the participants will receive the first questionnaire (pre-test). Once this questionnaire has been completed, a link to the app and the access code for the app will be provided. Participants will receive an invitation to complete the post-test after 10 days. Reminders to complete the questionnaire will follow after 2 and 4 days. All questionnaires are completed online.
  Interventions: Behavioral: Smartphone App

INTERVENTIONS:
Behavioral: Smartphone App — This intervention is a mobile app co-created with adolescents who have experienced suicidal thoughts. It is specifically designed for youth aged 12-17 and includes a Safety Plan, tools such as a HopeBox, and psychoeducational content for young people, their loved ones, and care providers. Furthermore, there is a 'Help' button, offering direct access to crisis support. Unlike existing apps for adults, this app is tailored to the developmental needs and lived experiences of adolescents. Access is restricted to study participants to ensure controlled evaluation.

SUMMARY:
There are currently very few evidence-based tools specifically designed to support children and adolescents experiencing suicidal thoughts. Digital interventions are increasingly used in suicide prevention and show promise in helping young people improve emotional regulation, coping skills, and manage suicidal thoughts and behaviors.

In Flanders, the app BackUp was developed in 2015 by VLESP to support adults with suicidal thoughts. Research showed that while the app led to a small, non-significant reduction in suicidal thoughts after one week, 70% of users found it helpful in daily life. A key feature of the app is the Safety Plan, based on cognitive behavioral therapy, which helps individuals identify coping strategies and sources of support. This approach has proven effective in reducing suicidal behavior and is also suitable for use with children and adolescents.

Despite these developments, there is still a need for a digital tool specifically tailored to young people. In 2023, the investigators launched a project to develop a new app in collaboration with youth care professionals, app developers, and adolescents with lived experience of suicidality. Their input ensures the app meets the needs and preferences of young users.

This study aims to evaluate the effectiveness and usability of the app through a pilot study involving adolescents aged 12-17 who are currently experiencing suicidal thoughts. Participants and their parents or guardians must provide informed consent before joining the study.

The evaluation includes online questionnaires completed before and after using the app. These questionnaires collect information on demographics, coping strategies, and the severity of suicidal thoughts and behaviors. The post-assessment also includes questions about user experience and satisfaction. No interviews are conducted; all data are collected digitally.

Participants are recruited through various channels and must meet specific inclusion criteria. After completing the initial questionnaire, they receive a code to access the app, ensuring that only study participants can use it.

DETAILED DESCRIPTION:
Research clearly shows that very few evidence-based tools or interventions exist specifically targeting suicidality in children and adolescents. Within suicide prevention there is increasing use of digital technology. Studies show that digital interventions aimed at suicidality in young people seem promising in terms of knowledge promotion, emotion regulation, development of coping skills and dealing with suicidal thoughts and behavior.

In Flanders in 2015, the app BackUp was developed by VLESP for adults struggling with suicidal thoughts. Research conducted by VLESP (reference number: 2015/0306) showed that use of the app led to a small but non-significant decrease in suicidal thoughts after one week. Moreover, 70% of users found the app useful in their daily lives. A key component of the app BackUp is the Safety Plan. Based on cognitive behavioral therapy, the Safety Plan aims to prevent suicidal behavior by establishing coping strategies and support resources. Since its introduction, the Safety Plan has been an integral part of standard care for suicidal individuals. The use of a Safety Plan has been shown to be effective in reducing suicidal behavior. In addition, research shows that it appears to be effective for use with children and adolescents.

However, there is a need for an app specifically aimed at young people, which they can use when they have suicidal thoughts. In 2023, the investigators initiated a project (EC code: ONZ-2024-0211) aimed at developing a mobile application through collaboration with professionals working in youth care, app developers, and co-creation with adolescents who have experienced suicidal thoughts. Throughout this process, young individuals with lived experience of suicidality actively contributed to the development of the app. This participatory approach ensures that the app is better aligned with their needs and help-seeking behaviors.

The next phase involves conducting an evaluation of the app. This evaluation seeks to gain deeper insights into its effectiveness and usability. To achieve this, the investigators will carry out a pilot study involving pre- and post-assessments with adolescents (aged 12-17) who are currently experiencing suicidal thoughts.

TThe pre- and post-assessments consist of online questionnaires completed by participants after both they and their parent or legal guardian have provided informed consent to participate in the study. During the pre-assessment, socio-demographic data are collected, along with information regarding suicide-related coping strategies and the severity of suicidal thoughts and behaviors. The post-assessment covers the same domains, supplemented with questions about user experience and satisfaction with the app.

No interviews are conducted as part of these assessments; all data are collected exclusively through online questionnaires.

Participants are specifically recruited for this study through various channels and must meet predefined inclusion criteria. Upon completion of the initial questionnaire, participants will receive an access code for the app. This procedure ensures that only adolescents who are explicitly enrolled in the study gain access to the app.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 through 17 years
* Currently experiencing suicidal thoughts (defined as a score of 1 or higher on the Suicidal Ideation Attributes Scale [SIDAS; Van Spijker et al., 2014])
* Access to the internet
* Possession of a smartphone
* Proficient in Dutch

Exclusion Criteria:

* Does not meet one or more of the inclusion criteria listed above

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of App Usage and User Experience | At post-test (Day 10 to day 14 after baseline assessment)
  The primary outcome of this study is to assess how young people use the app and their experience with its usability and perceived effectiveness. The evaluation focuses on identifying strengths and potential barriers within the target group to improve the app's accessibility and relevance. If participants have not completed the post-test questionnaire by Day 10, reminder messages are sent on Day 12 and Day 14.

SECONDARY OUTCOMES:
Suicide-Related Coping and Severity of Suicidal Thoughts and Behaviors | At Baseline (Day 0) and at Post-test (Day 10 to day 14 after baseline assessment)
  The secondary objective is to explore changes in suicide-related coping strategies and the severity of suicidal thoughts and behaviors. As this is a pilot study, the aim is not to demonstrate a clinically significant effect, but to assess the feasibility and applicability of the intervention. Findings may offer initial insights into which app components support adolescents in managing suicidal thoughts and inform future effectiveness studies. If participants have not completed the post-test questionnaire by Day 10, reminder messages are sent on Day 12 and Day 14 to encourage completion.

OTHER OUTCOMES:
Socio-demographic data | At Baseline (Day 0)
  Participants will be asked to provide basic demographic information, including gender identity, age, educational background, cultural background, sexual orientation, and any history of receiving mental health support.

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — University Ghent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided